CLINICAL TRIAL: NCT07046741
Title: Etat de Lieux de l'Allaitement Maternel Exclusif et Facteurs Prédictifs au CH de Martigues
Brief Title: Status Report on Exclusive Breastfeeding and Predictive Factors at Martigues Hospital
Acronym: EAME_FAP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Martigues (Other)
Responsible Party: Sponsor
Other Study IDs: CHMartigues
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Evaluate the Prevalence of Exclusive Breastfeeding at M0 (From the Birth of the Child) Within the Martigues CH; Breast Feeding Exclusive
Keywords: Breast Feeding; Infant Nutrition Disorders
MeSH Terms: conditions — Breast Feeding; Infant Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the prevalence of exclusive breastfeeding at M3 within the Martigues CH.

DETAILED DESCRIPTION:
After delivery, the investigating midwife or investigating pediatrician can go to the room where the new mother is installed to present the study to her. Once the patient consents, an information note will be given to her after signing a non-opposition.

The investigator or designated caregiver will produce the hetero-questionnaire in paper form to be completed depending on the patient's availability.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 and over
* Having given birth to a healthy child (or multiples) regardless of the number of weeks of amenorrhea
* Women practicing exclusive breastfeeding from the birth of the newborn
* Able to speak, read and understand French
* Having given oral consent

Exclusion Criteria:

* Minor mothers
* Refusal of consent
* Mothers wishing to practice artificial breastfeeding upon leaving the maternity ward will be excluded in M1 and M3
* Women who have changed their mind about exclusive breastfeeding during their maternity stay will be excluded

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women practicing exclusive breastfeeding from the birth of the newborn
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Rate of maternal breastfeeding at three month (M3) | up of 3 month
  Proportion of mothers that continue exclusive breastfeeding at 3 months at Martigues Hospital

SECONDARY OUTCOMES:
Rate of exclusive breastfeeding at 1 month (M1) | 1 month
  Proportion of mothers practicing exclusive breastfeeding at 1 month at Martigues Hospital

OTHER OUTCOMES:
Rate of exclusive breastfeeding at 3 months (M3) | 3 months
  Proportion of mothers practicing exclusive breastfeeding at 3 months at Martigues Hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Martigues, Martigues, Bouches du Rhone, France